CLINICAL TRIAL: NCT04686942
Title: Evaluation of Contrast Sonazoid-enhanced Ultrasound for the Detection of Colorectal Liver Metastases Less Than 2 cm
Brief Title: Sonazoid-enhanced Ultrasound for the Detection of Colorectal Liver Metastases Less Than 2 cm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yunfei Yuan, Professor, Sun Yat-sen University
Other Study IDs: Sonazoid001
Record Dates: First submitted 2020-12-20; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Liver Metastasis Colon Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before sonazoid: US detection liver metastases before sonazoid
- After sonazoid: US detection liver metastases after sonazoid
  Interventions: Diagnostic Test: After sonazoid

INTERVENTIONS:
Diagnostic Test: After sonazoid — 0.015ml/mg sonazoid enhanced US to detection of liver metastases.
  Groups: After sonazoid

SUMMARY:
Preoperative chemotherapy is often used for patients with colorectal cancer liver metastasis (CLM). Many small CLMs (<=2cm) may disappear after chemotherapy, while most of these are still alive. Ultrasonography (US) is a common imaging modality for the intraoperative detection tumor. Sonazoid is new echo-contrast agent, which is more stable and sensitive for detecting of small tumor. Investigators initially this prospective study to compare the detection performance before and after using sonazoid.

ELIGIBILITY:
Inclusion Criteria:

* Pathology confirmed colorectal adenocarcinoma
* One or more liver metastases less than 2 cm
* Multidisciplinary team recommend to perform preoperative chemotherapy
* Have baseline EOB-MR before chemotherapy

Exclusion Criteria:

* Could not fulfill the criteria of no evidence of disease (NED) after hepatic resection/ablation/radiotherapy
* With other malignancies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with one or more liver metastases lesions less than 2cm.
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
sensitive of detection tumor | 6 months
  Change of the sensitivity detection liver tumors when using sonazoid enhanced ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Yunfei Yuan, MD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided